CLINICAL TRIAL: NCT00576472
Title: Learning Impairments Among Survivors of Childhood Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MEMFX2; R01CA078957 (NIH); U01CA081445 (NIH); P30CA021765 (NIH)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2012-04-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2013-02

CONDITIONS: Acute Lymphoblastic Leukemia; Brain Tumors
Keywords: Brain Tumor, Acute Lymphoblastic Leukemia, Methylphenidate, Cognitive Late Effects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Brain Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — Please see detailed description for dosing information and study design.

SUMMARY:
Children surviving some types of cancer have a higher risk of developing learning problems after cancer treatment than do children who have not had cancer or its treatment. Cancer treatment may cause problems with learning, attention, and memory. The purpose of this study is to identify brain changes that may underlie learning problems in cancer survivors and investigate whether methylphenidate (a stimulant medication) may reduce these problems.

Subjects who have had treatment for acute lymphoblastic leukemia (ALL) or a brain tumor will be asked to take part in this research study. Siblings of some subjects will also be asked to take part, so that their results can be compared with those of children who have had cancer treatment. We hypothesize that children receiving more aggressive therapy will have lower white matter brain volumes and these volumes will be significantly lower than age-matched siblings. We also hypothesize that children who take methylphenidate will show improvements on teacher and parent report measures of attention and social skills.

DETAILED DESCRIPTION:
This study is a multi-phase, multi-site methylphenidate (MPH) trial in childhood cancer survivors. Study participants that meet inclusion and exclusion criteria are screened to ensure that they have adequate global cognitive functioning (IQ > 50) and have academic and attention difficulties that might be managed with MPH. Following the screening phase, qualifying participants take part in a two-day, in-clinic, double-blind, cross-over trial during which they receive MPH (0.6 mg/kg; maximum dose, 20 mg) and placebo (inert substance) in a randomly assigned order. Patients who do not have a significant adverse reaction during the two-day trial go on to participate in a randomized, double-blind, placebo-controlled, three-week home cross-over trial consisting of placebo, low-dose MPH (0.3 mg/kg; maximum dose, 10 mg bid), and moderate-dose MPH (0.6 mg/kg; maximum dose, 20 mg bid). Patients are then selected for participation in a 12-month open-label MPH trial if they show improvement over placebo on a parent and/or teacher rating of attention during the three-week home cross-over trial. The 12-month open-label MPH trial includes individually titrated MPH dosing to maximize clinical benefit, monthly monitoring of side effects and regular acquisition of parent and teacher ratings of attention and behavior. Laboratory measures of intellectual function, attention and memory are conducted at the end of the 12-month trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 to 18 years old.
* Active subject at St. Jude Children's Research Hospital, or is an age-matched sibling control subject.
* If a subject, received treatment for brain tumor or ALL with either radiation therapy and/or chemotherapy directed at the brain.
* If a subject, at least 12 months post-completion of antineoplastic therapies
* If a subject, no evidence of malignancy, or continuously stable disease since completion of therapy
* English as a primary language
* Informed consent

Exclusion Criteria:

* Glaucoma
* Patient or immediate family member with a history of Tourette's syndrome
* Current antidepressant, anxiolytic, antipsychotic or stimulant therapy
* History of substance abuse
* Recent history of uncontrolled seizures
* Uncorrected hypothyroidism
* Previously or currently randomized on COGRM1 intervention arm
* Previously diagnosed with ADHD, or, if a patient, diagnosed with ADHD prior to diagnosis of malignancy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 469 (Actual)
Dates: Start 2000-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Conklin, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Mulhern RK, Khan RB, Kaplan S, Helton S, Christensen R, Bonner M, Brown R, Xiong X, Wu S, Gururangan S, Reddick WE. Short-term efficacy of methylphenidate: a randomized, double-blind, placebo-controlled trial among survivors of childhood cancer. J Clin Oncol. 2004 Dec 1;22(23):4795-803. doi: 10.1200/JCO.2004.04.128. PMID 15570081
- [Background] Reddick WE, Shan ZY, Glass JO, Helton S, Xiong X, Wu S, Bonner MJ, Howard SC, Christensen R, Khan RB, Pui CH, Mulhern RK. Smaller white-matter volumes are associated with larger deficits in attention and learning among long-term survivors of acute lymphoblastic leukemia. Cancer. 2006 Feb 15;106(4):941-9. doi: 10.1002/cncr.21679. PMID 16411228
- [Background] Conklin HM, Khan RB, Reddick WE, Helton S, Brown R, Howard SC, Bonner M, Christensen R, Wu S, Xiong X, Mulhern RK. Acute neurocognitive response to methylphenidate among survivors of childhood cancer: a randomized, double-blind, cross-over trial. J Pediatr Psychol. 2007 Oct;32(9):1127-39. doi: 10.1093/jpepsy/jsm045. Epub 2007 Jun 14. PMID 17569711
- [Background] Reeves CB, Palmer S, Gross AM, Simonian SJ, Taylor L, Willingham E, Mulhern RK. Brief report: sluggish cognitive tempo among pediatric survivors of acute lymphoblastic leukemia. J Pediatr Psychol. 2007 Oct;32(9):1050-4. doi: 10.1093/jpepsy/jsm063. Epub 2007 Oct 12. PMID 17933846
- [Derived] Conklin HM, Lawford J, Jasper BW, Morris EB, Howard SC, Ogg SW, Wu S, Xiong X, Khan RB. Side effects of methylphenidate in childhood cancer survivors: a randomized placebo-controlled trial. Pediatrics. 2009 Jul;124(1):226-33. doi: 10.1542/peds.2008-1855. PMID 19564304
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 505 patients were enrolled from 3 institutions between January, 2000 and February, 2009. 91 siblings were enrolled as a control group.
Pre-assignment Details: Of 505 patients enrolled on the study, 36 were never assessed, and 469 participated in the initial screening. Of the 469 screened patients, 259 did not qualify for further medication phases, 75 qualified but refused to participate and 1 did not show for a scheduled appointment, leaving 134 patients to participate in the two-day MPH In-Lab Phase.
Groups:
- Mild Intensity: Intensity of prior CNS Therapy (systemic and/or intrathecal chemotherapy only)classified as mild.
- Moderate Intensity: Intensity of prior CNS Therapy (< 24 Gy CRT with or without systemic and/or intrathecal chemotherapy)classified as moderate.
- High Intensity: Intensity of prior CNS Therapy (>24 Gy CRT with or without systemic and/or intrathecal chemotherapy) classified as high.
- Screened/Didn't Qualify for Methylphenidate (MPH) In-Lab Phase: Of the 469 screened patients, 259 did not qualify for further medication phases, 75 qualified but refused to participate and 1 did not show for a scheduled appointment, leaving 134 patients to participate in the two-day Methylphenidate (MPH) In-Lab Phase.
- Group M/P: Group M/P (patients received oral Methylphenidate (MPH) and then an oral placebo)
- Group P/M: Group P/M (patients received oral placebo and then Methylphenidate (MPH))
- Completed MPH In-Lab Phase/Not Randomized for Cross Over Phase: Patients who completed the MPH in Lab Phase but were not randomized for the MPH Cross-Over Phase
- Placebo/Low Dose/Moderate Dose (PLM): The PLM group received a placebo on week one, low dose Methylphenidate (MPH) on week two, and a moderate dose of Methylphenidate (MPH) on week three.
- Placebo/Moderate Dose/Low Dose (PML): The PML group received a placebo on week one, moderate dose Methylphenidate (MPH) on week two, and a low dose of Methylphenidate (MPH) on week three.
- Low Dose/Moderate Dose/ Placebo (LMP): The LMP group received a low dose of Methylphenidate (MPH) on week one, a moderate dose of Methylphenidate (MPH) on week two, and a placebo on week three.
- Low Dose/Placebo/Moderate Dose (LPM): The LPM group received a low dose of Methylphenidate (MPH) on week one, a placebo on week two, and a moderate dose of Methylphenidate (MPH) on week three.
- Moderate Dose/Low Dose/Placebo (MLP): The MLP group received a moderate dose of Methylphenidate (MPH) on week one, a low dose of Methylphenidate (MPH) on week two, and a placebo on week three.
- Moderate Dose/Placebo/Low Dose (MPL): The MPL group received a moderate dose of Methylphenidate (MPH) on week one, a placebo on week two, and a low dose of Methylphenidate (MPH) on week three.
- Declined Methylphenidate (MPH) Home Maintenance Phase: Patients who completed the Methylphenidate (MPH) Cross Over Phase but chose to decline participation in the Methylphenidate (MPH) Home Maintenance Phase.
- Methylphenidate (MPH) Home Maintenance Phase: Methylphenidate (MPH) was administered for 12 months during the Methylphenidate (MPH) Home Maintenance Phase.
Period: Initial Screening
Arm/Group | Mild Intensity | Moderate Intensity | High Intensity | Screened/Didn't Qualify for Methylphenidate (MPH) In-Lab Phase | Group M/P | Group P/M | Completed MPH In-Lab Phase/Not Randomized for Cross Over Phase | Placebo/Low Dose/Moderate Dose (PLM) | Placebo/Moderate Dose/Low Dose (PML) | Low Dose/Moderate Dose/ Placebo (LMP) | Low Dose/Placebo/Moderate Dose (LPM) | Moderate Dose/Low Dose/Placebo (MLP) | Moderate Dose/Placebo/Low Dose (MPL) | Declined Methylphenidate (MPH) Home Maintenance Phase | Methylphenidate (MPH) Home Maintenance Phase
Started | 230 | 40 | 199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 230 | 40 | 199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MPH In-Lab Phase
Arm/Group | Mild Intensity | Moderate Intensity | High Intensity | Screened/Didn't Qualify for Methylphenidate (MPH) In-Lab Phase | Group M/P | Group P/M | Completed MPH In-Lab Phase/Not Randomized for Cross Over Phase | Placebo/Low Dose/Moderate Dose (PLM) | Placebo/Moderate Dose/Low Dose (PML) | Low Dose/Moderate Dose/ Placebo (LMP) | Low Dose/Placebo/Moderate Dose (LPM) | Moderate Dose/Low Dose/Placebo (MLP) | Moderate Dose/Placebo/Low Dose (MPL) | Declined Methylphenidate (MPH) Home Maintenance Phase | Methylphenidate (MPH) Home Maintenance Phase
Started | 0 (Group only associated with Screening phase.) | 0 (Group only associated with Screening phase.) | 0 (Group only associated with Screening phase.) | 335 | 67 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 67 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 335 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Declined participation in medication pha | 0 | 0 | 0 | 75 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patients did not qualify - IQ < 50 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No attention/academic problems | 0 | 0 | 0 | 245 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Psychiatric exclusion | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MPH Cross Over Phase
Arm/Group | Mild Intensity | Moderate Intensity | High Intensity | Screened/Didn't Qualify for Methylphenidate (MPH) In-Lab Phase | Group M/P | Group P/M | Completed MPH In-Lab Phase/Not Randomized for Cross Over Phase | Placebo/Low Dose/Moderate Dose (PLM) | Placebo/Moderate Dose/Low Dose (PML) | Low Dose/Moderate Dose/ Placebo (LMP) | Low Dose/Placebo/Moderate Dose (LPM) | Moderate Dose/Low Dose/Placebo (MLP) | Moderate Dose/Placebo/Low Dose (MPL) | Declined Methylphenidate (MPH) Home Maintenance Phase | Methylphenidate (MPH) Home Maintenance Phase
Started | 0 (Group not associated with MPH Cross-over phase.) | 0 (Group not associated with MPH Cross-over phase.) | 0 (Group not associated with MPH Cross-over phase.) | 0 (Group not associated with MPH Cross-over phase.) | 0 (Group not associated with MPH Cross-over phase.) | 0 (Group not associated with MPH Cross-over phase.) | 12 | 20 | 18 | 22 | 23 | 18 | 21 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 16 | 22 | 22 | 17 | 21 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible due to disease | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not complete cross over phase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Period: MPH Home Maintenance Phase
Arm/Group | Mild Intensity | Moderate Intensity | High Intensity | Screened/Didn't Qualify for Methylphenidate (MPH) In-Lab Phase | Group M/P | Group P/M | Completed MPH In-Lab Phase/Not Randomized for Cross Over Phase | Placebo/Low Dose/Moderate Dose (PLM) | Placebo/Moderate Dose/Low Dose (PML) | Low Dose/Moderate Dose/ Placebo (LMP) | Low Dose/Placebo/Moderate Dose (LPM) | Moderate Dose/Low Dose/Placebo (MLP) | Moderate Dose/Placebo/Low Dose (MPL) | Declined Methylphenidate (MPH) Home Maintenance Phase | Methylphenidate (MPH) Home Maintenance Phase
Started | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 0 (Group not associated with Home Maintenance Phase.) | 27 | 91
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 68
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 23
Not completed — Did not meet response criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0
Not completed — Declined to participate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Not completed — Insufficient data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Side effects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Medical reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Mild: Intensity of prior Central Nervous System radiation therapy was considered mild.
- Moderate: Intensity of prior Central Nervous System radiation therapy was considered moderate.
- High: Intensity of prior Central Nervous System radiation therapy was considered high.
- Not Randomized-In Lab Phase: Patients not randomized for the MPH in Lab Phase
- Group M/P: Group M/P (patients receive oral Methylphenidate (MPH) and then an oral placebo)
- Group P/M: Group P/M (patients receive oral placebo and ten Methylphenidate (MPH))
- Not Randomized-Cross Over: Patients who completed the MPH in Lab Phase but were not randomized for the MPH Cross Over Phase
- Placebo/Moderate Dose/Low Dose (PML): The PML group received a placebo on week one, moderate dose Methylphenidate (MPH) on week two, and a lose dose of Methylphenidate (MPH) on week three.
- Declined Home Maintenance Phase: Patients who completed the MPH Cross Over Phase but chose to decline participation in the Home Maintenance Phase.
- Home Maintenance Phase: Methylphenidate (MPH) was administered for 12 months during the duration of the Home Maintenance Phase.
- Total: Total of all reporting groups
Arm/Group | Mild | Moderate | High | Not Randomized-In Lab Phase | Group M/P | Group P/M | Not Randomized-Cross Over | Placebo/Low Dose/Moderate Dose (PLM) | Placebo/Moderate Dose/Low Dose (PML) | Low Dose/Moderate Dose/ Placebo (LMP) | Low Dose/Placebo/Moderate Dose (LPM) | Moderate Dose/Low Dose/Placebo (MLP) | Moderate Dose/Placebo/Low Dose (MPL) | Declined Home Maintenance Phase | Home Maintenance Phase | Total
Number analyzed (Participants) | 230 | 40 | 199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 469
Age, Customized [Number; unit: Participants]
  < 4 years of age | 113 | 23 | 51 |  |  |  |  |  |  |  |  |  |  |  |  | 187
  ≥ 4 years of age | 117 | 17 | 148 |  |  |  |  |  |  |  |  |  |  |  |  | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 16 | 90 |  |  |  |  |  |  |  |  |  |  |  |  | 204
  Male | 132 | 24 | 109 |  |  |  |  |  |  |  |  |  |  |  |  | 265
Disease Group [Number; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 216 | 39 | 3 |  |  |  |  |  |  |  |  |  |  |  |  | 258
  Brain Tumors (BT) | 14 | 1 | 196 |  |  |  |  |  |  |  |  |  |  |  |  | 211

OUTCOME MEASURES:

1. Primary Outcome: Brain White Matter Volume for Patients Versus Sibling Controls
Description: To compare the white matter volume of patients with those of sibling controls using MRI results captured between -1.8 and 42.36 months from study enrollment. Existing MRIs very close to enrollment were permissable for inclusion in this study.
Time Frame: Enrollment to evaluation of MRI, on average 12.8 months.
Population: Of the 505 patients enrolled, 106 did not have MRI acquired to measure brain volume, 16 were not evaluable: 6 had metal artifacts, 3 had motion artifacts, 1 had an acquisition error in MRI image, 4 had tumor on exam, and 2 had ischemic insults. 383 patients had evaluable MRI images. 67 of the 91 sibling controls had evaluable MRI images.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- Patients: Patients with evaluable MRIs.
- Siblings: Sibling controls with evaluable MRIs.
Arm/Group | Patients | Siblings
Number analyzed (Participants) | 383 | 67
percentage | 27 [26.5 to 27.5] | 30.3 [29.6 to 31]
Statistical Analysis 1: Comparison: Patients vs Siblings; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = -0.033, 95% CI 2-sided [-0.0452 to -0.0208], Standard Error of Mean 0.0062

2. Primary Outcome: Brain White Matter Volume for Patients With Acute Lymphoblastic Leukemia Versus Brain Tumors
Description: To compare the white matter volume of Acute Lymphoblastic Leukemia (ALL) patients with those of patients with malignant brain tumors using MRI results captured between -1.8 and 42.36 months from study enrollment. Existing MRIs very close to enrollment were permissable for inclusion in this study.
Time Frame: Enrollment to evaluation of MRI, on average 12.8 months.
Population: Of the 505 patients enrolled, 106 did not have MRI acquired to measure brain volume, 16 were not evaluable: 6 had metal artifacts, 3 had motion artifacts, 1 had an acquisition error in MRI image, 4 had tumor on exam, and 2 had ischemic insults. 383 patients had evaluable MRI images.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- Patients With ALL: Patients with Acute Lymphoblastic Leukemia (ALL) who had evaluable MRIs.
- Patients With Brain Tumors: Patients with brain tumors who had evaluable MRIs.
Arm/Group | Patients With ALL | Patients With Brain Tumors
Number analyzed (Participants) | 199 | 184
percentage | 28.4 [27.6 to 29.1] | 25.5 [25 to 26]
Statistical Analysis 1: Comparison: Patients With ALL vs Patients With Brain Tumors; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = 0.0285, 95% CI 2-sided [0.0190 to 0.0380], Standard Error of Mean 0.0046

3. Primary Outcome: Brain White Matter Volume for Treatment Intensity Groups and Sibling Controls
Description: To compare the white matter volume of patients by treatment intensity groups (mild, moderate, and high) and sibling controls using MRI results captured between -1.8 and 42.36 months from study enrollment. Existing MRIs very close to enrollment were permissable for inclusion in this study.
Time Frame: Enrollment to evaluation of MRI, on average 12.8 months.
Population: Of the 505 patients enrolled, 106 did not have MRI acquired to measure brain volume, 16 were not evaluable: 6 had metal artifacts, 3 had motion artifacts, 1 had an acquisition error in MRI image, 4 had tumor on exam, and 2 had ischemic insults. 383 patients had evaluable MRI images. 67 of the 91 sibling controls had an evaluable MRI image.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- Siblings: The sibling control group received no radiation therapy.
- Mild Treatment Intensity: Mildly intense central nervous system therapy (systemic and/or intrathecal chemotherapy only)
- Moderate Treatment Intensity: Moderately intense central nervous system therapy (<= 24 Gy CRT with or without systemic and/or intrathecal chemotherapy).
- High Treatment Intensity: High intensity central nervous system therapy (>24 Gy CRT with or without systemic and/or intrathecal chemotherapy.
Arm/Group | Siblings | Mild Treatment Intensity | Moderate Treatment Intensity | High Treatment Intensity
Number analyzed (Participants) | 67 | 173 | 34 | 176
percentage | 30.3 [29.6 to 31] | 28.8 [28 to 29.7] | 25.9 [24.3 to 27.5] | 25.4 [24.9 to 25.9]
Statistical Analysis 1: Comparison: Siblings vs Mild Treatment Intensity; Test type: Superiority or Other; p = 0.025, ANOVA; Mean Difference (Final Values) = 0.0144, 95% CI 2-sided [0.000204 to 0.0285], Standard Error of Mean 0.0064
Statistical Analysis 2: Comparison: Siblings vs Moderate Treatment Intensity; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = 0.0442, 95% CI 2-sided [0.0292 to 0.0591], Standard Error of Mean 0.0093
Statistical Analysis 3: Comparison: Siblings vs High Treatment Intensity; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = 0.0491, 95% CI 2-sided [0.0396 to 0.0586], Standard Error of Mean 0.0064
Statistical Analysis 4: Comparison: Mild Treatment Intensity vs Moderate Treatment Intensity; Test type: Superiority or Other; p = .0004, ANOVA; Mean Difference (Final Values) = 0.0298, 95% CI 2-sided [0.00974 to 0.0499], Standard Error of Mean 0.0083
Statistical Analysis 5: Comparison: Mild Treatment Intensity vs High Treatment Intensity; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = 0.0347, 95% CI 2-sided [0.0250 to 0.0445], Standard Error of Mean 0.0047
Statistical Analysis 6: Comparison: Moderate Treatment Intensity vs High Treatment Intensity; Test type: Superiority or Other; p = .552, ANOVA; Mean Difference (Final Values) = 0.00494, 95% CI 2-sided [-0.00865 to 0.0185], Standard Error of Mean 0.0083

4. Primary Outcome: Change From Methylphenidate (MPH) Home Maintenance Phase Baseline to Completion of Phase as Measured by Conners' Teacher Rating Scale (CTRS: ADHD T Score)
Description: The Conners' Teacher Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Twenty-eight questions are rated on a scale from 0 (not true at all) to 3 (very much true). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed prior to beginning the Methylphenidate (MPH) Home Maintenance Phase(baseline) and upon completion of the phase. Phase completion ranged between 11.44 and 24.36 months.
Time Frame: From beginning and at completion of Methylphenidate (MPH) Home Maintenance Phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 55 were screened at the beginning of the trial using the CTRS: ADHD T Score Questionnaire and 59 were screen at completion. 47 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 55 were screened at the beginning of the trial using the CTRS: ADHD T Questionnaire and 59 were screen at completion. 47 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 47
T-score | -7.17 [-11.0 to -3.3]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = .0005, ANOVA; Mean Difference (Final Values) = -7.17, 95% CI 2-sided [-11.0 to -3.3], Standard Error of Mean 1.93

5. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Conners' Teacher Rating Scale (CTRS: Cognitive Problem T Score)
Description: The Conners' Teacher Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Twenty-eight questions are rated on a scale from 0 (not true at all) to 3 (very much true). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and at completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 55 were screened at the beginning of the trial using the CTRS: ADHD T Score Questionnaire and 59 were screened at completion. 47 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 55 were screened at the beginning of the trial using the CTRS: Cognitive Problem T Score Questionnaire and 59 were screen at completion. 47 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 47
T-score | -3.34 [-6.5 to -0.1]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = 0.0413, ANOVA; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-6.5 to -0.1], Standard Error of Mean 1.59

6. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Conners' Parent Rating Scale (CPRS: ADHD T Score)
Description: The Conners' Teacher Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Twenty-seven questions are rated on a scale from 0 (not true at all) to 3 (very much true). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 and 24.36 months.
Time Frame: From beginning and at completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the CPRS: ADHD T Score Questionnaire and 68 were screen at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the CPRS: ADHD T Questionnaire and 68 were screen at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | -8.74 [-11.0 to -6.4]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = -8.74, 95% CI 2-sided [-11.0 to -6.4], Standard Error of Mean 1.20

7. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Conner's Parent Rating Scale (CPRS: Cognitive Problem T Score)
Description: The Conners' Teacher Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Twenty-seven questions are rated on a scale from 0 (not true at all) to 3 (very much true). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and at completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the CPRS: Cognitive Problem T Score Questionnaire and 68 were screened at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the CPRS: Cognitive Problem T Questionnaire and 68 were screen at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | -9.56 [-12.0 to -7.0]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = -9.56, 95% CI 2-sided [-12.0 to -7.0], Standard Error of Mean 1.3

8. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Social Skill Rating System (SSRS-P)
Description: The Social Skills Rating System- Parent Version (SSRS-P) is a parent rating scale of social behaviors in reference to typically developing children. Thirty eight questions are rated 0 (Never) to 3 (very often). The social skills score is norm-referenced with a mean of 100±15 where a higher score is indicative of better skills. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and at completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the Social Skills Rating System (SSRS-P) and 68 were screened at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the Social Skills Rating System and 68 were screened at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | 7.99 [4.4 to 11.6]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p < .0001, ANOVA; Mean Difference (Final Values) = 7.99, 95% CI 2-sided [4.4 to 11.6], Standard Error of Mean 1.81

9. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Wechsler Individual Achievement Test (WIAT) Reading: Composite Standard Score
Description: The Wechsler Individual Achievement Test is an examiner administered measure of academic skills. The Reading Composite consists of Basic Reading (single word reading) and Reading Comprehension. Raw scores are converted to standard scores with a mean of 100±15 where higher scores indicate better performance. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and at completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the Wechsler Individual Achievement Test (WIAT) REading: Composite Standard Score questionnaire and 68 were screened at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the WIAT Reading: Composite Standard Score System and 68 were screened at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | -0.21 [-2.3 to 1.9]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = .8425, ANOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-2.3 to 1.9], Standard Error of Mean 1.03

10. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Wechsler Individual Achievement Test (WIAT) Spelling: Standard Score
Description: The Wechsler Individual Achievement Test is an examiner administered measure of academic skills. The Spelling score assesses the child's ability to spell words to dictation. Raw scores are converted to standard scores with a mean of 100±15 where higher scores indicate better performance. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and after completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the Wechsler Individual Achievement Test (WIAT) Spelling: Standard Score System and 68 were screened at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the WIAT Spelling: Standard Score System and 68 were screened at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | -2.41 [-3.9 to -0.9]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = .0016, ANOVA; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-3.9 to -0.9], Standard Error of Mean 0.73

11. Primary Outcome: Change From Maintenance Phase Baseline to Completion of Phase as Measured by Wechsler Individual Achievement Test (WIAT) Math: Composite Standard Score
Description: The Wechsler Individual Achievement Test is an examiner administered measure of academic skills. The Math Composite score assesses the child's ability to solve calculation problems (Numerical Operations) and solve applied, word problems (Math Reasoning). Raw scores are converted to standard scores with a mean of 100±15 where higher scores indicate better performance. Assessments were performed prior to beginning the Home Therapy Phase (baseline) and upon completion of the phase. Phase completion ranged between 11.44 to 24.36 months
Time Frame: From beginning and after completion of home maintenance phase, on average 16.3 months.
Population: 118 patients began the MPH Home Maintenance Phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the Wechsler Individual Achievement Test (WIAT) Math: Composite Standard Score System. 68 were screened at completion. 68 patients were analyzed.
Measure: Mean (95% Confidence Interval); unit: T-score
Groups:
- Overall: 118 patients began the home maintenance phase of the trial. 68 completed the year long phase. 68 were screened at the beginning of the trial using the WIAT Math: Composite Standard Score System and 68 were screened at completion. 68 patients were screened at both the beginning and end of the home maintenance phase.
Arm/Group | Overall
Number analyzed (Participants) | 68
T-score | 0.22 [-1.9 to 2.3]
Statistical Analysis 1: Comparison: Overall; Test type: Superiority or Other; p = .8329, ANOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.9 to 2.3], Standard Error of Mean 1.04

12. Secondary Outcome: Best Weekly Score Measured by Conners' Parent Rating Scale (CPRS: ADHD T Score) During the 3-week Home Crossover Phase.
Description: The Conners' Teacher Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Twenty-seven questions are rated on a scale from 0 (not true at all) to 3 (very much true). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were done weekly during the 3-week Home Crossover Period with the best response being used as the measurement for the test.
Time Frame: weekly during 3-week home crossover phase
Population: There were 122 patients treated in the home crossover period. Some patients had missing treatments and outcome assessments. A crossover design was used for better efficiency of test and better precision of estimation.
Measure: Mean (95% Confidence Interval); unit: T score
Groups:
- Placebo: Patients assigned to the placebo group were randomly assigned to receive one of two arms: Group PLM received placebo during week one, low dose during week 2, and moderate dose during week 3; Group PML received placebo during week one, moderate dose during week 2, and low dose during week 3.
- Low Dose: Patients assigned to the Low Dose group were randomly assigned to receive one of two arms: Group LMP received low dose during week one, moderate dose during week 2, and placebo during week 3; Group LPM received low dose during week one, placebo during week 2, and moderate dose during week 3.
- Moderate Dose: Patients assigned to the Moderate Dose group were randomly assigned to receive one of two arms: Group MLP received moderate dose during week one, low dose during week 2, and placebo during week 3; Group MPL received moderate dose during week one, placebo during week 2, and low dose during week 3.
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
T score
  Oppositional T Score | 49.49 [39 to 89] | 50.87 [39 to 90] | 50.44 [39 to 88]
  Cognitive Problems/Inattention T Score | 55.64 [41 to 90] | 53.14 [41 to 87] | 51.72 [41 to 90]
  Hyperactivity T Score | 51.96 [42 to 88] | 51.14 [42 to 82] | 50.63 [42 to 90]
  Adhd T Score | 55.45 [25 to 90] | 53.08 [40 to 84] | 52.23 [40 to 90]

13. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Parent Rating Scale (CPRS) Cognitive Problem/Inattention Scale.
Description: The Conners' Parent Rating Scale- Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Three scales are reported: Cognitive Problems/Inattention (assesses the ability to learn at the same pace as peers, organize and complete work, and concentrate for sustained periods of time), Hyperactivity (assesses the ability to sit still to complete tasks, and impulsivity) and ADHD Index (assesses risk for ADHD disorder to be corroborated by other clinical information). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: 122 children began the Home Crossover Trial. 121 received all the placebo, 119 received all of the low dose, and 109 received all of the moderate dose.
Measure: Mean (Standard Error); unit: Estimated T Score
Groups:
- Placebo: Children qualifying for the 3-week, randomized Home MPH Crossover Trial will receive a combination of placebo, a low dose condition (0.3 mg/kg MPH; 10 mg maximum), and a moderate dose condition (0.6 mg/kg MPH; 20 mg maximum). There are six possible combinations of placebo (P), low dose MPH (LD), and moderate dose MPH (MD). Of the 122 children who began the Home Crossover Trial, 121 received the placebo. T Scores were estimated using a mixed model to account for carry-over effects. Mean and standard error were estimated by eliminating the effect of the carry-over from the directly measured mean.
- Low Dose: Children qualifying for the 3-week, randomized Home MPH Crossover Trial will receive a combination of placebo, a low dose condition (0.3 mg/kg MPH; 10 mg maximum), and a moderate dose condition (0.6 mg/kg MPH; 20 mg maximum). There are six possible combinations of placebo (P), low dose MPH (LD), and moderate dose MPH (MD). Of the 122 children who began the Home Crossover Trial, 119 received the low dose. T Scores were estimated using a mixed model to account for carry-over effects. Mean and standard error were estimated by eliminating the effect of the carry-over from the directly measured mean.
- Moderate Dose: Children qualifying for the 3-week, randomized Home MPH Crossover Trial will receive a combination of placebo, a low dose condition (0.3 mg/kg MPH; 10 mg maximum), and a moderate dose condition (0.6 mg/kg MPH; 20 mg maximum). There are six possible combinations of placebo (P), low dose MPH (LD), and moderate dose MPH (MD). Of the 122 children who began the Home Crossover Trial, 109 received the moderate dose. . T Scores were estimated using a mixed model to account for carry-over effects. Mean and standard error were estimated by eliminating the effect of the carry-over from the directly measured mean.
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 57.6595 (1.1335) | 54.6491 (1.0969) | 52.9854 (1.1368)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0077, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.1408, t-test, 2 sided

14. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Parent Rating Scale (CPRS) Hyperactivity Scale.
Description: as for outcome 13
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 54.2138 (1.0193) | 52.2771 (0.9899) | 51.5143 (1.0222)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0428, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0058, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.4258, t-test, 2 sided

15. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Parent Rating Scale (CPRS) ADHD Index.
Description: as for outcome 13
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 57.5805 (1.0861) | 54.4226 (1.0512) | 53.5317 (1.0893)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0035, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.4086, t-test, 2 sided

16. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Teacher Rating Scale (CTRS) Cognitive Problem/Inattention Scale.
Description: The Conners' Teacher Rating Scale-Revised (S) is a measure of the observed frequency of behaviors associated with ADHD. Three scales are reported: Cognitive Problems/Inattention (assesses the ability to learn at the same pace as peers, organize and complete work, and concentrate for sustained periods of time), Hyperactivity (assesses the ability to sit still to complete tasks, and impulsivity) and ADHD Index (assesses risk for ADHD disorder to be corroborated by other clinical information). Raw scores are converted to T scores using age and gender normative data. T scores have a mean of 50 ± 10 where higher scores are indicative of greater problems. Assessments were performed at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 62.7053 (1.0602) | 59.3272 (1.0368) | 59.6638 (1.0629)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.7007, t-test, 2 sided

17. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Teacher Rating Scale (CTRS) Hyperactivity Scale.
Description: as for outcome 16
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 55.7638 (1.1300) | 52.1765 (1.1034) | 52.6495 (1.1331)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0016, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.6237, t-test, 2 sided

18. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by The Conners' Teacher Rating Scale (CTRS) ADHD Index.
Description: as for outcome 16
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated T Score | 58.7691 (1.1050) | 54.7438 (1.0720) | 54.1974 (1.1084)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.6071, t-test, 2 sided

19. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by Social Skills Rating System - Parent (SSRS-P) - Social Skill.
Description: The SSRS assesses social skills for children and adolescents at preschool, elementary and secondary developmental levels. The SSRS is 40 to 57 items, depending on age, completed separately by parents (SSRS-P) and teachers (SSRS-T). Respondents rate the frequency of occurrence for each item ranging from 0 to 2 (0-never, 1-sometimes, 2-very often). The raw scores for the SSRS-P and SSRS-T Social Skills Scales and the SSRS-P and SSRS-T Problem Behaviors Scales have different ranges that are dependent upon age. Raw scores obtained from the SSRS Scales cannot be used to directly interpret social skills or problem behaviors as raw scores vary in meaning based on scale, informant form and developmental level. Raw scores are converted to standard scores with a mean of 100 ± 15. For the Social Skills Scale, a higher score is indicative of better social functioning, and for the Problem Behaviors Scale, a higher score is indicative of greater behavior problems.
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated Standard Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated Standard Score | 99.4412 (1.7590) | 101.5457 (1.7210) | 101.8999 (1.7632)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.1386, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0905, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.8039, t-test, 2 sided

20. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by Social Skills Rating System - Parent (SSRS-P) - Problem Behavior.
Description: as for outcome 19
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated Standard Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated Standard Score | 97.4890 (1.3408) | 97.0891 (1.3021) | 97.5709 (1.3446)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.7496, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.9489, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.7021, t-test, 2 sided

21. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by Social Skills Rating System - Teacher (SSRS-T) - Social Skill.
Description: as for outcome 19
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated Standard Score
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated Standard Score | 97.6171 (1.5035) | 100.6957 (1.4591) | 102.5281 (1.5012)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.0190, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.1622, t-test, 2 sided

22. Secondary Outcome: Effectiveness of MPH in Enhancing Classroom Attentiveness, Academic Productivity, and Social Behavior Measured by Social Skills Rating System - Teacher (SSRS-T) - Problem Behavior.
Description: as for outcome 19
Time Frame: Evaluated at the end of each medication week during the Home Therapy Phase- placebo, low dose and moderate dose weeks.
Population: as for outcome 13
Measure: Mean (Standard Error); unit: Estimated Standard Score
Groups:
- Moderate Dose: Children qualifying for the 3-week, randomized Home MPH Crossover Trial will receive a combination of placebo, a low dose condition (0.3 mg/kg MPH; 10 mg maximum), and a moderate dose condition (0.6 mg/kg MPH; 20 mg maximum). There are six possible combinations of placebo (P), low dose MPH (LD), and moderate dose MPH (MD). Of the 122 children who began the Home Crossover Trial, 109 received the moderate dose. T Scores were estimated using a mixed model to account for carry-over effects. Mean and standard error were estimated by eliminating the effect of the carry-over from the directly measured mean.
Arm/Group | Placebo | Low Dose | Moderate Dose
Number analyzed (Participants) | 121 | 119 | 109
Estimated Standard Score | 100.6084 (1.3671) | 98.6610 (1.3234) | 97.3103 (1.3661)
Statistical Analysis 1: Comparison: Placebo vs Low Dose; Test type: Superiority or Other; p = 0.1202, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Moderate Dose; Test type: Superiority or Other; p = 0.0103, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Dose vs Moderate Dose; Test type: Superiority or Other; p = 0.2831, t-test, 2 sided

23. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Sustained Attention, Reaction Time, and, Impulsivity Using Conner's Continuous Performance Test (CPT) for Omission Errors.
Description: Change in raw scores for the shortened version of the Conner's CPT from Baseline to Post-dose. The continuous performance test used during the in-lab trial was developed in house using SuperLab Pro v2.0 (Cedrus Corp., Phoenix, AZ). The test was modeled after Conners' CPT, but was shortened for ease of administration and evaluation of short-form sensitivity. The test is one-sixth the length of the Conners' CPT, lasting 2.33 min with 54 total targets and six nontargets (10% of trials). Similar to the Conners' CPT, the interstimulus intervals also varied by trial blocks with lengths of 1, 2, or 4 s. Omission errors are the raw score for the number of targets presented where the subject did not respond. Accordingly, the range for this variable is 0-54 with a higher score indicative of worse performance or problems with sustained attention.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: A mixed model was used to estimate the means of MPH and Placebo accounting for carry-over effects in the In-Lab crossover phase.
Measure: Mean (Standard Error); unit: Estimated raw score
Groups:
- MPH (Methylphenidate); Placebo; MPH Versus Placebo: Of the 469 screened patients, 259 did not qualify for further medication phases, 75 qualified but refused to participate and 1 did not show for a scheduled appointment, leaving 134 patients to participate in the two-day Methylphenidate (MPH) In-Lab Phase. 67 patients were assigned to the Group M/P sequence and 67 were assigned to the Group P/M sequence. Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We tested the difference in effects of MPH and placebo not the difference of two sequence groups.
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 129 | 129 | 129
Estimated raw score | 1.8889 (0.4923) | 1.6269 (0.4773) | 0.2620 (0.6857)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.7027, t-test, 2 sided

24. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Sustained Attention, Reaction Time, and, Impulsivity Using Conner's Continuous Performance Test (CPT) for Commission Errors.
Description: Change in raw scores for the shortened version of the Conner's CPT from Baseline to Post-dose. The continuous performance test used during the in-lab trial was developed in house using SuperLab Pro v2.0 (Cedrus Corp., Phoenix, AZ). The test was modeled after Conners' CPT, but was shortened for ease of administration and evaluation of short-form sensitivity. The test is one-sixth the length of the Conners' CPT, lasting 2.33 min with 54 total targets and six nontargets (10% of trials). Similar to the Conners' CPT, the interstimulus intervals also varied by trial blocks with lengths of 1, 2, or 4 s. Commission errors are the raw score for the numbers of nontargets presented where the subject incorrectly responded. Accordingly, the range for this variable is 0-6 with a higher score indicative of worse performance or impulsivity.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated raw score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 129 | 129 | 129
Estimated raw score | 3.6984 (0.2274) | 3.5970 (0.2205) | 0.1014 (0.3168)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.7493, t-test, 2 sided

25. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Sustained Attention, Reaction Time, and, Impulsivity Using Conner's Continuous Performance Test (CPT) for Hit Reaction Time.
Description: Change in raw scores for the shortened version of the Conner's CPT from Baseline to Post-dose. The continuous performance test used during the in-lab trial was developed in house using SuperLab Pro v2.0 (Cedrus Corp., Phoenix, AZ). The test was modeled after Conners' CPT, but was shortened for ease of administration and evaluation of short-form sensitivity. The test is one-sixth the length of the Conners' CPT, lasting 2.33 min with 54 total targets and six nontargets (10% of trials). Similar to the Conners' CPT, the interstimulus intervals also varied by trial blocks with lengths of 1, 2, or 4 s. Hit reaction time is average reaction time in milliseconds for all correct responses when targets were presented. There is no pre-defined range for reaction time; higher score is indicative of slower processing speed.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated raw score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 128 | 128 | 128
Estimated raw score | 350.0590 (10.1432) | 354.8515 (9.7573) | -4.7925 (14.0744)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.7339, t-test, 2 sided

26. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Sustained Attention, Reaction Time, and, Impulsivity Using Conner's Continuous Performance Test (CPT) for d' (Sensitivity).
Description: Change in raw scores for the shortened version of the Conner's CPT from Baseline to Post-dose. The continuous performance test used during the in-lab trial was developed in house using SuperLab Pro v2.0 (Cedrus Corp., Phoenix, AZ). The test was modeled after Conners' CPT, but was shortened for ease of administration and evaluation of short-form sensitivity. The test is one-sixth the length of the Conners' CPT, lasting 2.33 min with 54 total targets and six nontargets (10% of trials). Similar to the Conners' CPT, the interstimulus intervals also varied by trial blocks with lengths of 1, 2, or 4 s. D' and β are derived variables from signal detection theory. D' is a measure of sensitivity of a person to the signal or target; a higher score is indicative of better performance or better sustained attention. D' was calculated as z(hit) - z(commission). Z-scores were calculated using the NORMSINV function in Microsoft Excel.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated raw score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 119 | 118 | 118
Estimated raw score | 1.6809 (0.1632) | 1.7972 (0.1632) | -0.1163 (0.2307)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.6148, t-test, 2 sided

27. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Sustained Attention, Reaction Time, and, Impulsivity Using Conner's Continuous Performance Test (CPT) for Beta (Risk Taking).
Description: Change in raw scores for the shortened version of the Conner's CPT from Baseline to Post-dose. The continuous performance test used during the in-lab trial was developed in house using SuperLab Pro v2.0 (Cedrus Corp., Phoenix, AZ). The test was modeled after Conners' CPT, but was shortened for ease of administration and evaluation of short-form sensitivity. The test is one-sixth the length of the Conners' CPT, lasting 2.33 min with 54 total targets and six nontargets (10% of trials). Similar to the Conners' CPT, the interstimulus intervals also varied by trial blocks with lengths of 1, 2, or 4 s. D' and β are derived variables from signal detection theory. β is a measure of response tendency; higher scores indicate a more conservative response pattern. β was calculated using the formula = -d'*.5*(NORMSINV(hits)-NORMSINV(false alarms)). In the case where the false alarm rate = 0 or the hit rate = 1.0, we used the standard correction of 1/2N and 1- 1/2N, respectively.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated raw score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 121 | 123 | 121
Estimated raw score | 0.2300 (0.0320) | 0.2647 (0.0320) | -0.0346 (0.0453)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.4456, t-test, 2 sided

28. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Learning and Recall Using California Verbal Learning Test (CVLT) Over Five Learning Trials.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the California Verbal Learning Test (CVLT) to estimate the effectiveness of MPH on laboratory measures of learning and recall. CVLT Trials 1-5 have a mean T Score of 50 and Standard Deviation of 10.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 132 | 131 | 131
Estimated T Score | 44.6970 (1.6195) | 45.9403 (1.6074) | -1.2433 (2.2818)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.5866, t-test, 2 sided

29. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Learning and Recall Using California Verbal Learning Test (CVLT) for Short Delay Free Recall.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the California Verbal Learning Test (CVLT) to estimate the effectiveness of MPH on laboratory measures of learning and recall. CVLT Z Score for Short Delay Free Recall has a mean of 0 and a standard deviation of 1.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated Z Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 132 | 131 | 131
Estimated Z Score | -0.3636 (0.1449) | -0.3358 (0.1438) | -0.0278 (0.2041)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.8918, t-test, 2 sided

30. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Learning and Recall Using California Verbal Learning Test (CVLT) for Long Delay Free Recall.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the California Verbal Learning Test (CVLT) to estimate the effectiveness of MPH on laboratory measures of learning and recall. CVLT Z Score for Long Delay Free Recall has a mean of 0 and a standard deviation of 1.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated Z Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 131 | 131 | 131
Estimated Z Score | -0.3692 (0.1484) | -0.2090 (0.1462) | -0.1603 (0.2083)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.4427, t-test, 2 sided

31. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Interference, Impulsivity, Cognitive Flexibility, and Selective Attention Using the Stroop Word-Color Association Test (Stroop) for Word Naming Time.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the Stroop Word-Color Association Test (Stroop) to estimate the effectiveness of MPH on laboratory measures of interference, impulsivity, cognitive flexibility, and selective attention. Stroop T scores for Word Naming Time have a mean of 50 and a standard deviation of 10.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 126 | 126 | 126
Estimated T Score | 39.0156 (1.0095) | 37.8571 (1.0175) | 1.1585 (1.4333)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.4203, t-test, 2 sided

32. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Interference, Impulsivity, Cognitive Flexibility, and Selective Attention Using the Stroop Word-Color Association Test (Stroop) for Color Naming Time.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the Stroop Word-Color Association Test (Stroop) to estimate the effectiveness of MPH on laboratory measures of interference, impulsivity, cognitive flexibility, and selective attention. Stroop T scores for Color Naming Time have a mean of 50 and a standard deviation of 10.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 126 | 126 | 126
Estimated T Score | 40.7031 (1.0218) | 39.8889 (1.0299) | 0.8142 (1.4507)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.5754, t-test, 2 sided

33. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Interference, Impulsivity, Cognitive Flexibility, and Selective Attention Using the Stroop Word-Color Association Test (Stroop) for Ink Color Naming Time.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the Stroop Word-Color Association Test (Stroop) to estimate the effectiveness of MPH on laboratory measures of interference, impulsivity, cognitive flexibility, and selective attention. Stroop T scores for Ink Color Naming Time have a mean of 50 and a standard deviation of 10.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 126 | 126 | 126
Estimated T Score | 45.1094 (1.0327) | 41.7937 (1.0409) | 3.3157 (1.4662)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.0251, t-test, 2 sided

34. Secondary Outcome: Establish the Effectiveness of MPH on Laboratory Measures of Interference, Impulsivity, Cognitive Flexibility, and Selective Attention Using the Stroop Word-Color Association Test (Stroop) for Interference Score.
Description: Patients were randomized into two sequence groups: 1) P/M: placebo followed by MPH; 2) M/P: MPH followed by placebo. We are interested in testing the difference of effects of MPH and placebo, not in testing the difference of two sequence groups. We will use the Stroop Word-Color Association Test (Stroop) to estimate the effectiveness of MPH on laboratory measures of interference, impulsivity, cognitive flexibility, and selective attention. Stroop T scores for Interference Score have a mean of 50 and a standard deviation of 10.
Time Frame: Subjects were tested in both the drug and placebo groups before and after taking either MPH or placebo.
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Estimated T Score
Arm/Group | MPH (Methylphenidate) | Placebo | MPH Versus Placebo
Number analyzed (Participants) | 126 | 126 | 126
Estimated T Score | 52.6875 (0.8870) | 50.6349 (0.8940) | 2.0526 (1.2593)
Statistical Analysis 1: Comparison: MPH Versus Placebo; Test type: Superiority or Other; p = 0.1049, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the trial duration from January, 2000 through October, 2009.
Arm/Group | Mild | Moderate | High
Serious Adverse Events (participants affected / at risk) | 0/230 | 0/40 | 0/199
Other Adverse Events (participants affected / at risk) | 0/230 | 0/40 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes